CLINICAL TRIAL: NCT05998278
Title: Diagnostic Performance of a Individualized Reduced-Core Biopsy Strategy in Prostate Cancer: A Prospective, Randomized Controlled Study
Brief Title: Personalized Optimization of Systematic Prostate Biopsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022WSJK030
Record Dates: First submitted 2023-06-26; First posted 2023-08-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Prostate Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: They were randomly divided into two groups. One group received systematic biopsy. The other group received Targeted biopsy + personalized reduced-core biopsy .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group received targeted biopsy plus personalized systematic biopsy
  Interventions: Procedure: Personalized Optimization of Systematic Prostate Biopsy
- Control group (No Intervention): Control group received systematic biopsy

INTERVENTIONS:
Procedure: Personalized Optimization of Systematic Prostate Biopsy — Login the model based on our previous study (https://daringsky.shinyapps.io/prediction_v2/) allows for input of age, BMI, serum PSA, size and location of suspicious lesions, PIRADS - V2 score, and prostate volume to generate an individualized needle distribution map,then targeted biopsy combined personalized optimization of systematic prostate biopsy was performed.
  Arms: Experimental group

SUMMARY:
Targeted biopsy combined systematic biopsy is the gold standard for diagnosis of prostate cancer. Excessive cores in systematic biopsy increases the risk of puncture trauma， bleeding and infection. On the basis of establishing a model with DRS stratification to reduce the cores of systematic biopsy, we propose the (12 cores -x) model innovatively. We hope that through this prospective study to verify the efficacy of the model and provide patients with a new biopsy model with high accuracy and fewer complications.

In this study， patients with suspected prostate cancer were randomly divided into two groups. Experimental group received targeted biopsy combined personalized systematic biopsy, and the control group received systematic biopsy .The differences of the detection rate of Prostate cancer between the two groups were compared.

DETAILED DESCRIPTION:
In this study, patients with suspected prostate cancer were were enrolled at our institution, a public referral tertiary center. After written consent was obtained，Patients were randomly assigned to the intervention or control group in a 1:1 ratio by a research nurse who was not involved in the clinical study, using Computer-generated randomization method. Once the allocation was established, neither patients nor investigators, including the member of the study who collected the data related to infectious events later, were blinded. Prior to biopsy, the following patient characteristics were obtained: age, BMI, serum PSA levels, location and size of the region of interest, and PIRADS-V2 score. Biopsy was performed by an experienced urologist using standard transperineal technique. The patient was placed in the lithotomy position and underwent either general anesthesia or local anesthesia (15 ml of 5% lidocaine was injected into the prostate capsule and apex under ultrasound guidance after the ultrasound probe was inserted transrectally for local anesthesia). Patients assigned to the experimental group were informed of the personalized systematic biopsy combined with targeted biopsy using the (12 cores -x) model (https://daringsky.shinyapps.io/prediction_v2/)， and the control group received systematic biopsy. A biopsy core was obtained using an 18-gauge 25cm needle and a spring needle biopsy gun. The primary endpoint was the rate of prostate cancer diagnosis, including clinically significant cases. The secondary endpoints included pain scores and complications such as hematuria, perineal hematoma, urinary tract infection, and urinary retention.

An interim analysis is planned after approximately 50% of the target sample size has completed follow-up for the primary endpoint. The interim analysis aims to:

1. assess safety data to ensure participant protection, and
2. explore preliminary efficacy trends.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with lesions found on rectal examination with any PSA value;
2. Patients with abnormal lesions found on imaging with any PSA value;
3. PSA >10.0 ng.ml-1;
4. Patients with PSA of 4.0-10.0 ng.ml-1 and fPSA/tPSA < 0.16; (5 ) mpMRI was performed prior to biopsy and Prostate Imaging Reporting and Data System (PI-RADS V2.1) assessment category ≥3

(6) Willing to truthfully fill in the subject survey scale; (7) Willing to undergo follow-up; (8) The patient himself or his authorized immediate family member has signed the informed consent for clinical trial.

Exclusion Criteria:

1. previous biopsy cases;
2. Patients who have undergone prostate-related surgery, radiotherapy, or anti-androgen therapy;
3. Patients whopresented with severe hemorrhoids or rectal stenosis, rendering them intolerant to transrectal ultrasound
4. clotting disordersPatients with severe systemic diseases, such as cardiovascular and cerebrovascular disorders, are not appropriate candidates for surgical intervention.
5. unable to follow the plan.

Ages: 50 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 330 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The detection rate of clinically significant prostate cancer. | 3 months after biopsy
  According to the pathological results after biopsy, the detection rate of clinically significant prostate cancer (csPCa) was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenlin Chen, Principal Investigator — Department of Urology, Fujian Union Hospital, Fujian Medical University
Locations (1):
- Department of Urology, Fujian Union Hospital, Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen Z, Qu M, Shen X, Jiang S, Zhang W, Ji J, Wang Y, Zhang J, Chen Z, Lin L, Li M, Wu C, Gao X. Establishment of an Individualized Predictive Model to Reduce the Core Number for Systematic Prostate Biopsy: A Dual Center Study Based on Stratification of the Disease Risk Score. Front Oncol. 2022 Feb 14;11:831603. doi: 10.3389/fonc.2021.831603. eCollection 2021. PMID 35237503